CLINICAL TRIAL: NCT06591702
Title: Investigation of the Validity, Reliability, and Responsiveness of BETY-Biopsychosocial Questionnaire in Individuals with Chronic Kidney Disease, on Dialysis, and Kidney Transplantation
Brief Title: Investigation of the Validity, Reliability, and Responsiveness of BETY-BQ in Chronic Kidney Disease, on Dialysis, and Kidney Transplantation
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 24/097
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Disease(CKD); Chronic Kidney Disease Requiring Chronic Dialysis; Kidney Transplantation
Keywords: biopsychosocial model; validity and reliability; BETY-BQ; Chronic Kidney Disease; Kidney Transplantation; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire study — Questionnaire application
  Other Names: BETY-Biopsychosocial Questionnaire

SUMMARY:
A review of the literature has shown that Chronic Kidney Disease (CKD) is strongly associated with an increasing degree of psychosocial impact, such as depression and anxiety and a decrease in quality of life. Therefore, while determining the psychosocial aspects of the disease gains importance, it is reported that determining and evaluating the biopsychosocial characteristics may facilitate the disease management of individuals. Considering that CKD is associated with various comorbidities, psychosocial features, and symptom burden, it is interpreted that patient-reported outcome measures may support the complex management of these individuals. Routine collection and use of patient-reported outcome measures may provide valuable data for understanding the disease from both individual and community perspectives, with the potential to improve the quality of care and outcomes.

The Cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY) is an innovative exercise model based on physical exercise and an example of a biopsychosocial approach developed for patients with rheumatism. The BETY-Biopsychosocial Questionnaire (BETY-BQ) was created by repeated statistics of improvement characteristics reported by individuals who participated in BETY sessions for many years. The BETY-BQ holistically assesses many biopsychosocial characteristics of the person, such as pain, functionality, mood, sociability, sexuality, and sleep. Therefore, there is a need for scales that assess these symptoms holistically in chronic kidney disease. BETY-BQ can be envisaged as an assessment tool for interdisciplinary healthcare team members who want to evaluate the CKD population, including individuals on dialysis and kidney transplant recipients. Since the BETY-BQ can assess biopsychosocial characteristics quickly and its structure was created with the feedback of individuals with chronic diseases, it aimed to examine its validation in this disease group.

In this study, which investigators planned to contribute to this field, investigators aimed to investigate the validity, reliability, and sensitivity of BETY-BQ in individuals diagnosed with chronic kidney disease on dialysis and kidney transplantation.

ELIGIBILITY:
Individuals with chronic kidney disease:

Inclusion Criteria:

* Being diagnosed with chronic kidney disease
* To be over 18 years old
* Consent of the participant

Exclusion Criteria:

* Acute infection
* Being diagnosed with cancer

Individuals on dialysis:

Inclusion Criteria:

* Being a dialysis patient
* To be over 18 years old
* Consent of the participant

Exclusion Criteria:

* Acute infection
* Being diagnosed with cancer

Kidney transplant recipients:

Inclusion Criteria:

* To have had a kidney transplant
* To be over 18 years old
* Consent of the participant

Exclusion Criteria:

* Acute infection
* Being diagnosed with cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | Three months
  The biopsychosocial status is evaluated through questions about pain, functionality, mood, sociability, sexuality, and sleep. Each question has 30 items, with scores ranging from 0 to 120, categorized as follows: 0 (never), 1 (yes rarely), 2 (yes sometimes), 3 (yes often), and 4 (yes always). Higher scores reflect a poorer biopsychosocial status.

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale | Three months
  The Hospital Anxiety and Depression Scale (HADS) comprises 14 items, with 7 items assessing anxiety and the other 7 evaluating depression. Each item is scored on a scale of 0 to 3, resulting in a total score ranging from 0 to 21. Higher scores indicate more severe levels of anxiety and depression.
Kidney Disease and Quality of Life™ (KDQOL™-36) | Three months
  The 36-item scale includes three specific dimensions: symptoms/problems, burden of kidney disease and effects of kidney disease, and physical component and mental component components derived from SF12. The scale, which consists of 5 sub-dimensions, is scored between 0-100. Higher scores indicate better health-related quality of life.
Clinical Frailty Scale | Three months
  A scale that can be easily administered in most clinical settings and is scored from 1 (very fit) to 9 (terminally ill) about fitness, active illness, activities of daily living, and cognition. The assessment is based on the subjective judgment of a clinician.
Frail Scale | Three months
  The FRAIL scale is based on a table of self-reported fatigue, mobility, strength, weight loss, and comorbidities. Each item is scored between 0-1, totaling 5 points. A high score indicates a high level of frailty.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals